CLINICAL TRIAL: NCT01302431
Title: An Exploratory Randomized Controlled Trial of a Manualized, Nurse-led, Telephone Intervention Support Service for Support Persons of People With Multiple Sclerosis
Brief Title: Nurse-Led Manualized Telephone Support Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Margarita Corry, Research fellow, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NLTSI
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Multiple Sclerosis
Keywords: experimental; intervention; nurse-led; nurse specialist; multiple sclerosis; support of caregivers
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nurse-Led Manualised Telephone support (Experimental): Participants assigned to this arm of the study will receive 4 nurse-led telephone support calls over a three month time-frame
  Interventions: Other: Manualised nurse-led telephone support
- Usual care (No Intervention): Participants randomised to this arm of the study will receive their usual care which comprises caregivers calling nurse specialists when they needs advice and support

INTERVENTIONS:
Other: Manualised nurse-led telephone support — The manualised nurse-led telephone support intervention is designed to provide proactive support and enable caregivers of people with multiple sclerosis manage problems encountered with caregiving
  Arms: Nurse-Led Manualised Telephone support

SUMMARY:
The primary aim of this study is to determine if a manual based telephone intervention support service for people who support people with Multiple Sclerosis (PwMS), initiated by nurse specialists who provide care to PwMS, has a positive impact on the lives of PwMS and their support persons. For support persons this impact is determined by measurable support person/carer self-efficacy and preparedness to care, burden, quality of life, service utilization and satisfaction with the support service. For PwMS this is determined by their qualitative experience of the type of care they receive from their carer. A secondary aim is to determine the possible economic benefits of the introduction of such an intervention nationally. A support person is the person nominated by the PwMS as the person who provides the most support or physical assistance to a person with MS who is not a paid service provider.

DETAILED DESCRIPTION:
The negative impact of caregiving on caregivers of People with Multiple Sclerosis (PwMS) has been well documented (Corry & While, 2008). Outside of scheduled health care contacts, caregivers usually make contact with nurse specialists when in distress or in crisis situations. Nurses specialising in MS have specialised knowledge in caring for PwMS and their caregivers and the management of symptoms of MS, and are well positioned to provide specialist advice, information and referral. Much of the unique support given to caregivers of PwMS by MS nurses in Ireland is undocumented so that their impact upon patient and carer outcomes is unknown.

The well-being of caregivers of PwMS is crucial with limited budgets resulting in increased reliance upon caregivers to provide ongoing support for PwMS. Health care professionals need to prioritise health promotion, information giving and pro-active management of situations among caregivers of PwMS if the deleterious effects of care-giving on the PwMS and their caregivers are to be minimised and poor health avoided.

A search of the literature revealed that no published studies exist on the use of telephone support interventions for caregivers of PwMS. The extent to which telephone support interventions have been used in an attempt to support caregivers is evident from the number of studies found on carer telephone support across a number of illnesses (n=29). The range of care recipients, research designs and objectives for the studies make it difficult to draw definitive conclusions regarding particular outcomes and interventions. However, positive findings include feeling supported (Bank et al. 2006, Stewart et al. 2001), feeling empowered (Wilkes et al. 2004; Stewart et al. 2001) and reduced carer burden (Bormann et al. 2009; Tremont et al. 2008; Stewart et al. 2001).

The positive findings from the studies on telephone support interventions, along with the current use of carer telephone contact with NSMS when in crisis, suggest that a nurse specialist proactive approach to problem management, information and advice giving has potential for positive outcomes for caregivers of PwMS.

For the purpose of this study a carer is defined as a person who provides the most support or physical assistance to a PwMS, and who is not a paid service provider.

ELIGIBILITY:
Inclusion Criteria:

PwMS:

* People who have a diagnosis of Multiple Sclerosis and are > 18 years of age.
* PwMS who nominate a caregiver.

Caregivers:

* Informal caregivers of PwMS who do not have a serious mental health problem.

Nurses: Nurse Specialists caring for PwMS and who agree to take part in the study.

Exclusion Criteria:

For PwMS:

* PwMS who cannot nominate a caregiver
* PwMS who are already engaged in similar research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2011-04; Primary Completion 2013-10 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Support person/caregiver Self-efficacy | 3 months
  This outcome measures support person/caregiver self-efficacy for obtaining respite and self-efficacy in problem solving

SECONDARY OUTCOMES:
Support person/caregiver preparedness to care | 3 months
  This outcome measure measures how well support persons/caregivers feel prepared to care for a PwMS

CONTACTS AND LOCATIONS:
Locations (2):
- Ireland (2):
  - Site 1, Dublin
  - Dublin

REFERENCES:
- [Background] Tremont G, Davis JD, Bishop DS, Fortinsky RH. Telephone-Delivered Psychosocial Intervention Reduces Burden in Dementia Caregivers. Dementia (London). 2008;7(4):503-520. doi: 10.1177/1471301208096632. PMID 20228893
- [Background] Stewart MJ, Hart G, Mann K, Jackson S, Langille L, Reidy M. Telephone support group intervention for persons with hemophilia and HIV/AIDS and family caregivers. Int J Nurs Stud. 2001 Apr;38(2):209-25. doi: 10.1016/s0020-7489(00)00035-3. PMID 11223062
- [Background] Bormann J, Warren KA, Regalbuto L, Glaser D, Kelly A, Schnack J, Hinton L. A spiritually based caregiver intervention with telephone delivery for family caregivers of veterans with dementia. Fam Community Health. 2009 Oct-Dec;32(4):345-53. doi: 10.1097/FCH.0b013e3181b91fd6. PMID 19752637
- [Background] Bank AL, Arguelles S, Rubert M, Eisdorfer C, Czaja SJ. The value of telephone support groups among ethnically diverse caregivers of persons with dementia. Gerontologist. 2006 Feb;46(1):134-8. doi: 10.1093/geront/46.1.134. PMID 16452294
- [Background] Corry M, While A. The needs of carers of people with multiple sclerosis: a literature review. Scand J Caring Sci. 2009 Sep;23(3):569-88. doi: 10.1111/j.1471-6712.2008.00645.x. Epub 2008 Dec 9. PMID 19077062